CLINICAL TRIAL: NCT04037709
Title: Efficacy of Photodynamic Therapy and Scraping in Patients With Gingivitis Predisposed by Fixed Orthodontic Appliances: Randomized, Controlled, Double-blind, Split-mouth Study
Brief Title: Photodynamic Therapy in Patients With Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Anna Carolina Ratto Tempestini Horliana, PhD, clinical professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PDT
Record Dates: First submitted 2019-07-24; First posted 2019-07-30 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2020-01

CONDITIONS: Gingivitis; Orthodontic Appliance Complication; Photodynamic Therapy
MeSH Terms: conditions — Gingivitis | interventions — Tooth Exfoliation; Root Planing; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Intervention Model Description: Patients will have their mouth divided into two groups: Control group (n = 17) - Scaling and Root Planing (SRP) + PDT placebo and Experimental group (n = 17) - SRP + PDT.
Who Masked: Participant, Investigator
Masking Description: Only the researcher responsible for conducting the treatments (who will open the randomized envelopes) will know which treatment is assigned to each patient. The identification of each group will only be revealed by this researcher after statistical analysis of the data for all those involved in the study. Therefore, the researcher responsible for data collection, the microbiologist and the statistician will be blind regarding the treatments assigned to the groups. The patient will also be blind to the type of treatment performed since the periodontal treatment will be identical in both groups and treatment with PDT will be simulated in the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scaling and root planing (SRP) + PDT placebo (Placebo Comparator): 17 patients will receive periodontal treatment (scaling and root planing - SRP) with the ultrasound. The SRP will be done in one session. SRP will be performed by only one experienced researcher. Periodontal reassessment will be performed after 30 days.
  The PDT placebo wil be done using an agent with the same vehicle as that of the methylene blue to mimic irrigation with the photosensitizer; the laser will be switched off at the time of application.
  Interventions: Procedure: scaling and root planing (SRP) + PDT placebo
- scaling and root planing (SRP) + PDT (Experimental): 17 patients will receive the same scaling and root planing treatment that placebo group.
  However the PDT will be done only on one side of the mouth using methylene blue 0.005% - Chimiolux 5, DMC - purified water and methylene blue.The red laser diode (λ = 660 nm) will be applied with an output power of 100mW . The laser head will be positioned in direct contact with the pseudo periodontal pocket.
  Interventions: Procedure: scaling and root planing (SRP) + PDT

INTERVENTIONS:
Procedure: scaling and root planing (SRP) + PDT placebo — Patientes will receive periodontal treatment (scaling and root planing - SRP) with the ultrasound. The SRP will be done in one session. The PDT placebo wil be done using an agent with the same vehicle as that of the methylene blue to mimic irrigation with the photosensitizer; the laser will be switched off at the time of application.
  Arms: scaling and root planing (SRP) + PDT placebo
Procedure: scaling and root planing (SRP) + PDT — patients will receive the same scaling and root planing treatment that placebo group.However the PDT will be done only on one side of mouth using methylene blue 0.005% .The red laser diode (λ = 660 nm) will be applied with an output power of 100mW . The laser head will be positioned in direct contact with the pseudo periodontal pockets.
  Arms: scaling and root planing (SRP) + PDT

SUMMARY:
The hypothesis to be tested in this study is whether photodynamic therapy (PDT) could favor the decontamination of these areas, as the photosensitizer and light are capable of reaching areas that these instruments have difficulty accessing. In other words, the objective of this study is to evaluate the impact of PDT as an adjuvant treatment to scaling, considering clinical immunoregulatory in patients with gingivitis with the predisposing factor of the use of a fixed orthodontic appliance. A randomized, controlled, double-blind, split-mouth clinical study will include 17 patients. Patients will have their mouth divided into two groups: Control group (n = 17) - Scaling and Root Planing (SRP) + PDT placebo and Experimental group (n = 17) - SRP + PDT. In G2 will be used methylene blue 0.005%, λ = 660nm, 9J (joule) per inflamed site, irradiance = 3.5W / cm (watts/centimeter), radiant exposure = 318J / cm2. In G1 and G2 the scaling will be performed with the aid of the ultrasound. All participants will receive oral hygiene guidance (OHG) after to the end of the study. The clinical periodontal data to be analyzed: plaque index (PI), gingival index (GI) and probing depth (PD) and clinical level of insertion (CLI) by means of a periodontal probe. Crevicular fluid will be collected (from 8 pre-determined sites) for analysis of the IL-6 (interleukin), IL-1β, IL-8, TNF-α (tumor necrosis factor) and IL-10 cytokines, using the ELISA method.

DETAILED DESCRIPTION:
It is known that the presence of orthodontic brackets predisposes for a change in both the quantity and quality of the biofilm, due to the challenge of brushing adequately. The sites are difficult to access with a toothbrush and periodontal curette, worsening inflammation. In addition, gingival growth is frequently associated with poor hygiene. The hypothesis to be tested in this study is whether photodynamic therapy (PDT) could favor the decontamination of these areas, as the photosensitizer and light are capable of reaching areas that these instruments have difficulty accessing. In other words, the objective of this study is to evaluate the impact of PDT as an adjuvant treatment to scaling, considering clinical and immunoregulatory parameters in patients with gingivitis with the predisposing factor of the use of a fixed orthodontic appliance. A randomized, controlled, double-blind, split-mouth clinical study will include 17 patients, both genders, having used the fixed appliance for more than 12 months, with gingivitis present. Patients will have their mouth divided into two groups: Control group (n = 17) - Scaling and Root Planing (SRP) + PDT placebo and Experimental group (n = 17) - SRP + PDT. In G2 methylene blue 0.005%, λ = 660nm, 9J (joule) per inflamed site, irradiance = 3.5W/ cm, radiant exposure = 318J/ cm2. In G1 and G2 the scaling will be performed with the aid of the ultrasound. All participants will receive oral hygiene guidance (OHG) after to the end of the study. The clinical periodontal data to be analyzed: plaque index (PI), gingival index (GI) and probing depth (PD) and clinical level of insertion (CLI) by means of a periodontal probe. Crevicular fluid will be collected (from 8 pre-determined sites) for analysis of the IL-6, IL-1β, IL-8, TNF-α and IL-10 cyttokines, using the ELISA method. All analysis will be realized using the baseline (T0) and (T1) 30 days after treatment. If sample distribution is normal, the Student T-test will be used to compare the measurement of continuous and dependent variables. If it is not normal, the Mann-Whitney test will be used. The data will be presented in terms of ± PD and the value of p will be defined as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* healthy participants (negative medical history),
* of both genders,
* aged 10 to 30 years,
* with gingivitis induced by dental biofilm,
* predisposed by the use of a fixed orthodontic appliance, according to the classification of 2018

Exclusion Criteria:

* participants with maxillary and mandibular deformities,
* periodontitis,
* oral lesions and who have used antibiotics for less than 3 months,
* those who have used non-steroidal anti-inflammatory drugs and continuous corticosteroid therapy for less than 3 months,
* who have been using mouthwash in the past 3 months.
* Participants who have modifying factors for periodontal disease, such as diabetics, immunosuppressive smokers (cyclosporine), anticonvulsants (phenytoin), calcium channel blockers (nifedipine) and pregnant and lactating women as well as those who are HIV positive, or have Hepatitis B or C. - Patients who require prophylactic antibiotic therapy for periodontal treatment - who have had periodontal treatment in the last 6 months.
* Patients who have non-biofilm-induced gum disease.
* Patients who for some reason during the study have to initiate the use of the medicines and mouthwashes mentioned above or acquire a disease that is a modifying factor for periodontal disease or become pregnant.
* Patients who do not wish to remain part of the study may drop out whenever they wish.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Gingival bleeding index | through study completion on average of one year
  The periodontal probe will be inserted at all predetermined sites at the gingival margin of all teeth, 30 seconds will be waited and, at the smallest sign of bleeding, the presence or absence of bleeding will be noted. Gingival bleeding will be evaluated at 4 sites (mesiobuccal, distobuccal, mesiolingual, distolingual.The gingival Index will be presented in a percentage (%). The result will be based on the ratio of total sites to sites affected. Results will be considered indicative of gingivitis with ≥ 10% bleeding . It will be assessed at baseline and 30 days after treatment.

SECONDARY OUTCOMES:
Clinical probing depth (PD) | through study completion on average of one year
  Will be done by a calibrated evaluator using a periodontal probe marked in millimeters (North Carolina University periodontal probe, UNC-15 (Hu-FriedyTM): all teeth (except third molars) will be evaluated at 4 sites (mesiobuccal, distobuccal, mesiolingual, distolingual) using the aforementioned parameters.
  The Northe Carolina University periodontal probe will be insert in the gingival sulcus. Probing depths to be evaluated in millimeters (mm) from the base of the periodontal pocket to the free gingival margin. It will be assesed at baseline and 30 days after treatment.
Evaluation of crevicular fluid cytokines IL-6, IL-1β, and IL-10, | through study completion on average of one year
  Evaluation of cytokines IL-6, IL-1β, , and IL-10, will be done via the ELISA. The paper cones will be inserted at regions with gingivitis and gingival hyperplasia (pseudo pocket) until resistance be felt. The cone will remain in this position for 30 seconds. If there is blood contamination a new cone will be used after 90 seconds. Eight cones must be collected, one for each site. The cones will be placed in a 1.5ml microcentrifuge tube and stored at -80 °C. It will be assesed at baseline and 30 days after treatment;

OTHER OUTCOMES:
Visible plaque index (PI) | through study completion on average of one year
  Will be visualy evalueted before of probing depht, using the following score of visible supragingival plaque:
  Presence = 1 Absence = 0 It will be assessed at baseline and 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Anna Carolina R Horliana, Phd, Principal Investigator — Nove de Julho University
Locations (1):
- Anna Carolina R.T. Horliana, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schalch TO, Palmieri M, Longo PL, Braz-Silva PH, Tortamano IP, Michel-Crosato E, Mayer MPA, Jorge WA, Bussadori SK, Pavani C, Negreiros RM, Horliana ACRT. Evaluation of photodynamic therapy in pericoronitis: Protocol of randomized, controlled, double-blind study. Medicine (Baltimore). 2019 Apr;98(17):e15312. doi: 10.1097/MD.0000000000015312. PMID 31027098
- [Result] Gomez C, Abellan R, Palma JC. Efficacy of photodynamic therapy vs ultrasonic scaler for preventing gingival inflammation and white spot lesions during orthodontic treatment. Photodiagnosis Photodyn Ther. 2018 Dec;24:377-383. doi: 10.1016/j.pdpdt.2018.11.001. Epub 2018 Nov 3. PMID 30399455
- [Result] Chapple ILC, Mealey BL, Van Dyke TE, Bartold PM, Dommisch H, Eickholz P, Geisinger ML, Genco RJ, Glogauer M, Goldstein M, Griffin TJ, Holmstrup P, Johnson GK, Kapila Y, Lang NP, Meyle J, Murakami S, Plemons J, Romito GA, Shapira L, Tatakis DN, Teughels W, Trombelli L, Walter C, Wimmer G, Xenoudi P, Yoshie H. Periodontal health and gingival diseases and conditions on an intact and a reduced periodontium: Consensus report of workgroup 1 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S74-S84. doi: 10.1002/JPER.17-0719. PMID 29926944
- [Derived] Rosa EP, Murakami-Malaquias-Silva F, Schalch TO, Teixeira DB, Horliana RF, Tortamano A, Tortamano IP, Buscariolo IA, Longo PL, Negreiros RM, Bussadori SK, Motta LJ, Horliana ACRT. Efficacy of photodynamic therapy and periodontal treatment in patients with gingivitis and fixed orthodontic appliances: Protocol of randomized, controlled, double-blind study. Medicine (Baltimore). 2020 Apr;99(14):e19429. doi: 10.1097/MD.0000000000019429. PMID 32243363